CLINICAL TRIAL: NCT05492500
Title: A PHASE 2, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, 4-ARM STUDY TO INVESTIGATE SYMPTOMS, FUNCTION, HEALTH-RELATED QUALITY OF LIFE AND SAFETY WITH REPEATED SUBCUTANEOUS ADMINISTRATION OF PONSEGROMAB VERSUS PLACEBO IN ADULT PARTICIPANTS WITH HEART FAILURE
Brief Title: A Study of Ponsegromab in People With Heart Failure
Acronym: GARDEN TIMI 74
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following a prespecified interim analysis, and in consultation with the independent Data Monitoring Committee, the Sponsor terminated the study
Sponsor: Pfizer (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: C3651011; 2023-509747-27-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-07-25; First posted 2022-08-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; N-terminal pro-B type natriuretic peptide; Kansas City Cardiomyopathy Questionnaire; Patient's Global Impression of Severity; Patient's Global Impression of Change; Patient Reported Outcome Measurement Information System; Growth differentiation factor 15; New York Heart Association
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: In the main cohort (Cohort A), ponsegromab will be administered at low, medium and high doses every 4 weeks by subcutaneous injections for a total of 6 doses. Participants will be randomized to 1 of the 3 doses of ponsegromab or placebo.
  In optional Cohort C, ponsegromab will be administered at low doses every 4 weeks by subcutaneous injections for a total of 6 doses. Participants will be randomized to the low dose of ponsegromab or placebo.
  In optional Cohort D, ponsegromab will be administered at high doses every 4 weeks by subcutaneous injections for a total of 6 doses. Participants will be randomized to the high dose of ponsegromab or placebo.
  In a separate open-label, PK cohort (Cohort B), ponsegromab will be administered at low, medium and high doses every 4 weeks by subcutaneous injections for a total of 4 doses. Participants will be randomized to 1 of the 3 doses of ponsegromab. There is no placebo in the open-label, PK cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the main cohort (Cohort A), Cohort C and Cohort D, investigators, sponsor, participants and other site staff will be blinded to participants' assigned study intervention, including the site staff assigned to prepare and administer the study intervention. Pharmacists and site personnel will be blinded to study intervention versus placebo within each study arm.
  The separate PK cohort (Cohort B) will be open-label and study treatment will be prepared and administered as per treatment assignment by qualified personnel. There is no blinding in the open-label, PK cohort (Cohort B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Main cohort (Cohort A): ponsegromab low dose (Experimental): Participants will receive a low dose Q4W SC
  Interventions: Drug: Main cohort (Cohort A): Ponsegromab low dose
- Main cohort (Cohort A): ponsegromab medium dose (Experimental): Participants will receive a medium dose Q4W SC
  Interventions: Drug: Main cohort (Cohort A): Ponsegromab medium dose
- Main cohort (Cohort A): ponsegromab high dose (Experimental): Participants will receive a high dose Q4W SC
  Interventions: Drug: Main cohort (Cohort A): ponsegromab high dose
- Main cohort (Cohort A): placebo (Placebo Comparator): matched placebo
  Interventions: Other: Main cohort (Cohort A): Matched placebo
- Open-label, PK Cohort (Cohort B): ponsegromab low dose (Experimental): Participants will receive a low dose Q4W SC
  Interventions: Drug: Open-label, PK Cohort (Cohort B): ponsegromab low dose
- Open-label, PK Cohort (Cohort B): ponsegromab medium dose (Experimental): Participants will receive a medium dose Q4W SC
  Interventions: Drug: Open-label, PK Cohort (Cohort B): ponsegromab medium dose
- Open-label, PK Cohort (Cohort B): ponsegromab high dose (Experimental): Participants will receive a high dose Q4W SC
  Interventions: Drug: Open-label, PK Cohort (Cohort B): ponsegromab high dose
- Optional Cohort C: ponsegromab low dose (Experimental): Participants will receive a low dose Q4W SC
  Interventions: Drug: Optional Cohort C: Ponsegromab low dose
- Optional Cohort C: placebo (Placebo Comparator): matched placebo
  Interventions: Other: Optional Cohort C: Matched placebo
- Optional Cohort D: ponsegromab high dose (Experimental): Participants will receive a high dose Q4W SC
  Interventions: Drug: Optional Cohort D: Ponsegromab high dose
- Optional Cohort D: placebo (Placebo Comparator): matched placebo
  Interventions: Other: Optional Cohort D: Matched placebo

INTERVENTIONS:
Drug: Main cohort (Cohort A): Ponsegromab low dose — Ponsegromab low dose subcutaneous injection
  Other Names: PF-06946860 low dose
  Arms: Main cohort (Cohort A): ponsegromab low dose
Drug: Main cohort (Cohort A): Ponsegromab medium dose — Ponsegromab medium dose subcutaneous injection
  Other Names: PF-06946860 medium dose
  Arms: Main cohort (Cohort A): ponsegromab medium dose
Drug: Main cohort (Cohort A): ponsegromab high dose — Ponsegromab high dose subcutaneous injection
  Other Names: PF-06946860 high dose
  Arms: Main cohort (Cohort A): ponsegromab high dose
Other: Main cohort (Cohort A): Matched placebo — Matched placebo subcutaneous injection
  Other Names: Placebo
  Arms: Main cohort (Cohort A): placebo
Drug: Open-label, PK Cohort (Cohort B): ponsegromab low dose — ponsegromab low dose subcutaneous injection
  Other Names: PF-06946860 low dose
  Arms: Open-label, PK Cohort (Cohort B): ponsegromab low dose
Drug: Open-label, PK Cohort (Cohort B): ponsegromab medium dose — Ponsegromab medium dose subcutaneous injection
  Other Names: PF-06946860 medium dose
  Arms: Open-label, PK Cohort (Cohort B): ponsegromab medium dose
Drug: Open-label, PK Cohort (Cohort B): ponsegromab high dose — Ponsegromab high dose subcutaneous injection
  Other Names: PF-06946860 high dose
  Arms: Open-label, PK Cohort (Cohort B): ponsegromab high dose
Drug: Optional Cohort C: Ponsegromab low dose — Ponsegromab low dose subcutaneous injection
  Other Names: PF-06946860 low dose
  Arms: Optional Cohort C: ponsegromab low dose
Other: Optional Cohort C: Matched placebo — Matched placebo subcutaneous injection
  Other Names: Placebo
  Arms: Optional Cohort C: placebo
Drug: Optional Cohort D: Ponsegromab high dose — Ponsegromab high dose subcutaneous injection
  Other Names: PF-06946860 high dose
  Arms: Optional Cohort D: ponsegromab high dose
Other: Optional Cohort D: Matched placebo — Matched placebo subcutaneous injection
  Other Names: Placebo
  Arms: Optional Cohort D: placebo

SUMMARY:
The primary purpose of this clinical trial is to compare the effects of study medicine (Ponsegromab/PF-06946860) with a placebo (an injection that looks like the study medicine but does not contain the active medicine) to find out if the study medicine is better than the placebo (an injection that looks like the study medicine but does not contain the active medicine) for treatment of symptoms related to heart failure. Participants will not know which treatment group they are assigned to. Most participants in this study will receive the study medicine or placebo by shots under the skin every four weeks. People may be able to participate in this study if they have heart failure. Participants will take part in this study for about 9 months. During this time participants will visit the study clinic once a month.

A separate PK cohort within this clinical trial will receive open-label study medicine (Ponsegromab/PF-06946860) only. Participants in this open-label, PK cohort will not receive placebo. These participants will receive the study medicine by shots under the skin every four weeks. People may be able to participate in this study cohort if they also have heart failure. Participants will take part in the open-label, PK cohort for about 7 months.

DETAILED DESCRIPTION:
The primary purpose of this study is to assess the effect of repeated subcutaneous administration of ponsegromab (PF-06946860) compared to placebo on frequency, severity, and burden of symptoms as well as physical limitations in participants with heart failure and different ranges of circulating GDF-15 concentrations. The study will also assess the safety, tolerability, PK, PD, and immunogenicity of ponsegromab.

A separate, open-label, PK cohort, with more frequent PK and GDF-15 collection after single and multiple subcutaneous administration of ponsegromab (PF-06946860), will be enrolled at certain sites to facilitate a more comprehensive assessment of PK characteristics and PK/PD relationship for GDF-15 in participants with heart failure and elevated circulating GDF-15 concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older

  -. Clinical evidence of HF with each of the following criteria:
  1. LVEF <50% on most recent measurement, within 12 months of screening. Note: An assessment of LVEF in the prior 12 months is not required in situations where LVEF has been persistently <50% on prior assessments obtained at least 3 months apart (including the most recent measurement).
  2. NYHA class II-IV at screening.
  3. NT-proBNP ≥400 pg/mL at screening (Note: Does not apply to open-label, PK Cohort [Cohort B]).
* Serum GDF-15 concentration ≥2000 pg/mL at screening.
* Cohort D only: Serum GDF-15 concentration <2000 pg/mL at screening.
* KCCQ-23 CSS <75 at screening (Note: Does not apply to open-label, PK Cohort [Cohort B]).
* Evidence of cachexia or fatigue or functional impairment, as demonstrated by at least one of the following at screening (Note: Does not apply to open-label, PK Cohort [Cohort B]):

  1. Non-edematous unintentional weight loss ≥5% in the last 6 months or current BMI <20 kg/m2, associated with subjective fatigue or anorexia; or
  2. Fatigue at least 3 times per week AND at least moderately bothersome fatigue in the past 2 weeks based on the KCCQ-23 administered at screening; or
  3. A score of <60 on the Physical Limitations Domain of the KCCQ 23 administered at screening.

Exclusion Criteria:

* Acute decompensated HF within 1 month prior to Screening Visit 1 or during the screening period.
* Implantation of a cardiac resynchronization therapy device or valve repair or replacement within 3 months prior to randomization or intent to do so during the trial.

For the open-label, PK cohort (Cohort B) only: implantation of a cardiac resynchronization therapy device more than 1 month prior to randomization is permitted.

* History of heart transplantation, currently listed for heart transplant, current/planned mechanical circulatory support, or current/planned use of intravenous inotropes (eg, dobutamine, milrinone).
* Acute coronary syndrome within 1 month prior to randomization.
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) within 3 months prior to randomization or intent to undergo coronary revascularization during the trial.

For the open-label, PK cohort (Cohort B) only: coronary revascularization more than 1 month prior to randomization is permitted.

* Untreated indication for an implantable cardiac defibrillator or pacemaker to treat a cardiac rhythm abnormality (ie, tachyarrhythmia or bradyarrhythmia).
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives (whichever is longer) preceding the first dose of study intervention used in this study. Treatment with an investigational biologic agent within 6 months or 5 half-lives (whichever is longer) of Day 1.
* Previous exposure to ponsegromab in a prior clinical study.
* Renal disease requiring ongoing dialysis.
* Cirrhosis with evidence of portal hypertension not due to HF, or the following LFT abnormalities at the time of screening, confirmed by a repeat test if deemed necessary: AST or ALT level ≥ 3 x ULN, or total bilirubin level ≥ 2 x ULN (unless history of Gilbert's syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Main cohort (Cohort A): Change from baseline in Kansas City Cardiomyopathy Questionnaire 23 Clinical Summary Score | baseline, 22 weeks
  To compare the effect of high dose ponsegromab versus placebo, on heart failure disease-specific health status in participants with HF and elevated serum GDF-15 concentrations

SECONDARY OUTCOMES:
Main cohort (Cohort A): Change from baseline in Kansas City Cardiomyopathy Questionnaire 23 Overall Summary Score | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific overall health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Change from baseline in Kansas City Cardiomyopathy Questionnaire 23 Total Symptom Score | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific overall health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Change from baseline in Kansas City Cardiomyopathy Questionnaire 23 physical limitations domain | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific overall health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Responses as defined by a ≥5 point increase from baseline in Kansas City Cardiomyopathy Questionnaire 23 Clinical Summary Score | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Responses as defined by a ≥5 point increase from baseline in Overall Summary Score | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Responses as defined by a ≥5 point increase from baseline in Total Symptom Score | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Responses as defined by a ≥5 point increase from baseline in physical limitation | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on HF disease-specific health status in participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Change from baseline in 6-Minute Walk Distance | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on the physical function of participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A): Change from baseline in PROMIS-Fatigue 7a which will be completed by study participants on an electronic device, so as to compare the effect of ponsegromab versus placebo on fatigue as reported by participants with HF | baseline, 22 weeks
  To compare the effect of ponsegromab versus placebo on fatigue reported by participants with HF and elevated serum GDF-15 concentrations
Main cohort (Cohort A)/Cohort C/Cohort D: Incidence of treatment-emergent adverse events | 32 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Main cohort (Cohort A)/Cohort C/Cohort D: Incidence of treatment-emergent serious adverse events | 32 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Main cohort (Cohort A)/Cohort C/Cohort D: Incidence of abnormal laboratory results | 32 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Main cohort (Cohort A)/Cohort C/Cohort D: Incidence of abnormal vital signs | 32 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Open-Label, PK Cohort (Cohort B): Incidence of treatment-emergent adverse events | 22 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Open-Label, PK Cohort (Cohort B): Incidence of treatment-emergent serious adverse events | 22 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Open-Label, PK Cohort (Cohort B): Incidence of abnormal laboratory results | 22 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF
Open-Label, PK Cohort (Cohort B): Incidence of abnormal vital signs | 22 weeks
  To describe the safety and tolerability of ponsegromab in participants with HF

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (121):
- United States (22):
  - Eastern shore Research Institute LLC, Fairhope, Alabama
  - Keck Medical Center of USC, Los Angeles, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University School of Medicine-Grady Campus, Atlanta, Georgia
  - Chicago Medical Research, Hazel Crest, Illinois
  - Reid Physician Associates, Richmond, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Traverse Heart & Vascular, Traverse City, Michigan
  - M Health Fairview Clinics and Surgery Center, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Investigational Drug Services, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center-East Bank, Minneapolis, Minnesota
  - University of Minnesota/Lillehei Clinical Research Unit, Minneapolis, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in St. Louis Center for Outpatient Health (COH), St Louis, Missouri
  - Washington University in St. Louis Center for Advanced Medicine (CAM), St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Clinical and Translational Research Center, Chapel Hill, North Carolina
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Texas Health Heart & Vascular Specialist (THHVS) #18760, Dallas, Texas
- Australia (5):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Core Research Group, Brisbane, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Canada (17):
  - Fraser Clinical Trials Inc, New Westminster, British Columbia
  - QEII Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Saul Vizel Professional Medicine Corporation dba Vizel Cardiac Research, Cambridge, Ontario
  - University Hospital - London Health Sciences Centre, London, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Private Practice - Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Corcare, Toronto, Ontario
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - Community Care Building, Winchester, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski, Rimouski, Quebec
  - CardioVasc HR Inc, Saint-Jean-sur-Richelieu, Quebec
  - Centre intégré de santé et de services sociaux de Lanaudière - Hopital Pierre-Le Gardeur., Terrebonne, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
- China (11):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - China-Japan Union Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Tianjin People' s Hospital, Tianjin, Tianjin Municipality
  - Peking University First Hospital, Beijing
- Czechia (6):
  - EDUMED - Jaroměř, Jaroměř, Náchod
  - Institut Klinicke a Experimentalni Mediciny, Prague, Praha 4
  - Fakultni Nemocnice u sv. Anny v Brne, Brno, South Moravian
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Ustredni vojenska nemocnice, Prague
- Germany (5):
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt am Main, Hesse
  - Universitätsmedizin Göttingen - Georg-August-Universität, Göttingen, Lower Saxony
  - Herz - und Diabeteszentrum Nordrhein - Westfalen, Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
- Hungary (8):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Private Practice - Dr. Lakatos Ferenc, Békéscsaba, Bekes County
  - TaNa Med, Mosonmagyaróvár, Győr-Moson-Sopron
  - Medifarma 98 Kft, Nyíregyháza, Nyíregyháza
  - Somogy Vármegyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Dél-Pesti Centrumkórház Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Kanizsai Dorottya Korhaz, Nagykanizsa
- Japan (10):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - National Hospital Organization Saitama Hospital, Wako, Saitama
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Osaka General Medical Center, Osaka
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - Kardio Brynow, Katowice, Silesian Voivodeship
  - Miejski Szpital Zespolony w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz
  - Polsko Amerykanskie Kliniki Serca, Tychy
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego Centralny Szpital Kliniczny, Warsaw
- Spain (17):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Región de
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (12):
  - Wycombe General Hospital, High Wycombe, Buckinghamshire
  - Ninewells Hospital and Medical School, Dundee, Dundee CITY
  - St. George's Hospital, London, England and Wales
  - Northwick Park Hospital, Harrow, London, CITY of
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Barnet Hospital, Barnet
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Golden Jubilee National Hospital, Clydebank
  - Lincoln County Hospital, Lincoln
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Northern General Hospital, Sheffield
  - University Hospital of North Tees, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651011